CLINICAL TRIAL: NCT02067520
Title: Intrathecal (IT) Hydromorphone for Cesarean Section (C/S): A Dose Finding Study
Brief Title: Intrathecal Hydromorphone for Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 13D.611
Record Dates: First submitted 2014-01-30; First posted 2014-02-20 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Pain
Keywords: Post C/S pain relief
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- IT hydromorphone dose (Other): dose response study
  Interventions: Drug: intrathecal hydromorphone (IT hydromorphone)

INTERVENTIONS:
Drug: intrathecal hydromorphone (IT hydromorphone)

SUMMARY:
Introduction:

Cesarean section (C/S) is usually performed under spinal with preservative free morphine for pain relief, but the investigators have a severe shortage of this formulation of morphine. Hydromorphone is a narcotic which acts peripherally and centrally to decrease pain. It has been used in spinals for postoperative pain relief and in pain pumps for relief of chronic pain. No randomized controlled studies have evaluated intrathecal (IT) hydromorphone for post C/S pain.

Methods:

This is a randomized double-blind controlled trial utilizing the up-down sequential allocation method1,2 to find the best dose of IT hydromorphone that provides pain relief following C/S. Patients will be given a morphine PCA pump for additional pain relief. Our first patient will receive 200 mcg of IT hydromorphone. Pain, nausea, and itching will be evaluated at 4, 8, 12 and 24 hours following the C/S via numeric rating scales; vomiting and morphine use per hour will be recorded. Success will be a median morphine usage of less than or equal to 1mg/hour in the following 16 hours. If a success, the next patient will be given 10 mcg less IT hydromorphone; if a failure, she will receive 10 mcg more. The study will end after 5 successes.

Objective:

The primary objective is to find the optimal dose of IT hydromorphone for pain relief following C/S. The secondary objectives are to define the incidence and severity of hydromorphone's side effects and determine the duration of analgesia.

DETAILED DESCRIPTION:
SpecificAims Cesarean section (C/S) is usually performed under spinal anesthesia with preservative free morphine added for pain relief, but currently the investigators have a severe shortage of this formulation of morphine. Hydromorphone is a narcotic which has been used in spinals for acute postoperative pain relief and in pain pumps for relief of chronic pain. The investigators hypothesize that a dose between 25 and 200 mcg of IT hydromorphone will provide pain relief for at least 16 hours following C/S, with the need for minimal rescue medication, and therefore may be a reasonable alternative to IT morphine.

Background and Significance Cesarean section is usually performed under spinal anesthesia using bupivacaine. Intrathecal preservative free morphine is often added to decrease postoperative pain for 12-24 hours with only the need for minor rescue medication (a significant intravenous and oral opioid sparing effect). This allows earlier mobilization and interaction with family/infant of these hypercoagulable patients. With the critical shortage of this formulation of morphine, we must find an alternative medication. Hydromorphone is a narcotic which acts peripherally and centrally to decrease pain. It has been used in spinal anesthetics for acute postoperative pain relief and in pain pumps for relief of chronic pain. Currently hydromorphone is not approved for intrathecal administration by the FDA, but pain practitioners commonly prescribe hydromorphone for intrathecal pumps and have so for years. The most recent Poly Analgesic Consensus Conference (PACC) of 2012 included IT hydromorphone as an acceptable opioid for chronic use. Its inclusion for the management of neuropathic and nociceptive pain infers hydromorphone's relative neurologic safety, as it is used in much higher doses than for cesarean section. The investigators reviewed the literature to learn if IT hydromorphone has been used for post C/S pain relief, and if so, at what dose. A retrospective chart review comparing IT hydromorphone to fentanyl after C/S and a case report of IT hydromorphone for a repeat C/S were all the investigators found.3,4 No randomized controlled studies exist.

Our study will find the optimal dose of IT hydromorphone for pain relief following cesarean section as well as delineate the incidence and severity of side effects and how long the drug lasts. This information is critical as no other viable alternatives currently exist to replace IT morphine in this capacity.

Preliminary Studies/Progress Report

The spinal anesthetic including the IT hydromorphone will be performed by a competent anesthesia resident or attending (residents on the obstetric anesthesia service, the principal investigator, or one of the co-investigators). Our C/S rate is about 31% of 2100 deliveries per year and most (>80%) are done under spinal.

Research Design and Methods

This is a randomized double-blind controlled trial utilizing the up-down sequential allocation method (continual reassessment)1,2 to find the best dose of IT hydromorphone that provides pain relief following C/S. Spinal anesthetic containing the specified dose of IT hydromorphone will be administered in the OR by the anesthesia resident or attending.

After consent is obtained, the first patient will be assigned to a dose of 200 mcg of IT hydromorphone. Although the dose of IT hydromorphone equivalent to that of IT morphine for post cesarean section pain is not known, some sources suggest that 50 - 100 mcg of IT hydromorphone may be similar to 100 - 200 mcg of IT morphine5-8. After preliminary observations using varying doses of IT hydromorphone for post C/S analgesia, the investigators observed that average and median morphine consumption in the following 16 hours was not markedly decreased until a dose of 200 mcg IT hydromorphone was reached (40 observational patients to date, no increased side effects). The investigators now use this dose routinely on labor and delivery so the investigators have chosen this as a starting dose. The spinal anesthetic will also include 15mg of hyperbaric bupivacaine. All patients will be provided with a morphine patient controlled analgesia (PCA) pump in the post-anesthesia care unit (PACU) for additional pain relief. At 4, 8, 12 and 24 hours following the C/S, the patient will rate her pain, degree of nausea, and itching with verbal numeric rating scales, (pain: 0 - 10, nausea and itching: 0 - 5) and the investigators will record the incidence of vomiting. These verbal numeric rating scales are commonly used at Thomas Jefferson for any patient using IV PCA pumps for postoperative pain. The investigators will also obtain a (validated) "quality of recovery scale" from each patient. Standard nursing orders include monitoring respiratory rate every 1 hour for 6 hours, then every 2 hours for 6 hours, for signs of respiratory depression, use of pulse oximetry, and administration of naloxone if needed. These orders are currently standard for all patients receiving IT preservative free morphine and are in an order set in Jeff Chart. The PCA pump will be queried the next day to evaluate the number of attempts and actual use of morphine in the first 16 hours postoperatively. The data will be compiled and analyzed by our statistician. Success will be defined as a median dose of less than or equal to 1mg/hour of morphine usage in the following 16 postoperative hours. If a patient is determined to be a success, the next patient will be assigned to a dose of IT hydromorphone that is 10 mcg less than the previous patient. (If the first patient is a success, the second patient will receive 190 mcg of IT hydromorphone). If a patient is deemed a failure, the next patient will receive a dose of IT hydromorphone that is 10 mcg higher than the previous patient. (If the first patient is a failure, the second patient will receive 210 mcg of IT hydromorphone). Our goal is to stop the study when the investigators get 5 points of success using the lowest concentration of IT hydromorphone resulting in a median dose of less than or equal to 1mg/hr of morphine consumption in the 16 hours post-operatively.

Statistical Methods This is a randomized double-blind controlled trial utilizing the up-down sequential allocation method of Dixon and Massey.1,2 On the basis of previous non-probability sequential dosing studies with binary outcomes (success vs failure), the investigators estimate on enrolling 40-50 patients.9-11 Using the referenced studies, the investigators estimate a minimum of 10 independent negative-positive up-and-down deflections in the study. Our goal is to stop the study when the investigators get 5 points of success using the lowest concentration of IT hydromorphone resulting in less than or equal to 1mg/hr of morphine consumption for 16 hours post-operatively.

All data will be analyzed using the Statistical Package for the Social Sciences (SPSS software, Version 21.0 (IBM Corporation). The continuous data will be reported as mean ± standard deviation (SD). Tests of significance include the t test for independent samples, Wilcoxon rank-sum test for non-parametric data and Chi-square or Fisher's exact test for frequency count data. Repeated measurements (pain scores, nausea scores) will be analyzed by repeated measure analysis of variance where normally distributed, with further paired comparisons at each time interval performed using the t-test. A P value < 0.05 will be considered significant. A dose response curve will also be created to determine the effective dose in 95% of patients (ED95) and effective dose in 50% of patients (ED50) for the patient population.

1. The investigators would like to enroll at least 40 - 50 patients as needed.
2. PCA pump attempts and usage for 16 hours, pain medication adjuncts used, verbal numeric rating scores for nausea, itching and pain, incidence of vomiting, and respiratory rate (recorded every one hour) will be obtained.
3. The patient will be approached if she meets inclusion criteria when she is admitted to the labor floor on the morning of her scheduled C/S. The study will be explained to her, the possible risks, benefits, and alternatives will be discussed, she will be given the opportunity to ask questions and if she agrees, the consent will be signed. The dose of IT hydromorphone will be determined and made up by our statistician physician. The spinal anesthetic will be administered to the patient in the operating room and the C/S will proceed as usual. Data will be collected over the next 16 hours according to the above research design.
4. Risks of any narcotic medication include analgesia, drowsiness, mental clouding, changes in mood, euphoria or dysphoria, respiratory depression, cough suppression, decreased gastrointestinal motility, nausea, vomiting, increased cerebrospinal fluid pressure, increased biliary pressure, pinpoint constriction of the pupils, increased parasympathetic activity and transient hyperglycemia. There is also the risk that the study drug is ineffective at controlling post C/S pain.
5. Standard nursing orders will include monitoring respiratory rate every 1 hour for 6 hours, then every 2 hours for 6 hours, for signs of respiratory depression, use of pulse oximetry, and administration of naloxone if needed. These orders are currently standard for all patients receiving IT preservative free morphine and are in an order set in Jeff Chart. They allow early recognition of and/or minimize the risk of respiratory depression should it occur. Also, the dosages the investigators will use are well below documented safe doses of this drug for the IT route. All patients will be provided with a morphine patient controlled analgesia (PCA) pump in the postanesthesia care unit (PACU) for additional pain relief whether or not the study drug is effective.
6. Potential benefit of the study is pain relief in the postoperative period following C/S (Our usual medication is currently unavailable or in critically limited supply).
7. The side effect profiles for our standard drug, IT morphine and the study drug IT hydromorphone are similar. Delayed respiratory depression and itching are more notable with IT morphine than described with IT hydromorphone so this may be beneficial. The duration of action of IT hydromorphone may not be as long as that of IT morphine.

This study poses minimal risk. This is a dose finding study. The dosages the investigators will use are well below documented safe doses of this drug for the IT route.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing a primary or repeat elective, scheduled C/S who are not yet in labor will be approached for inclusion in the study

Exclusion Criteria:

* Patient refusal,
* Age less than 18 years
* Onset of labor
* Current opioid abuse
* Use of methadone maintenance for previous opioid abuse
* Allergy to hydromorphone
* Contraindication to spinal anesthesia
* Inability to obtain a spinal anesthetic
* Language other than English or if unable to understand use of a PCA pump will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to find the optimal dose of IT hydromorphone for pain relief following C/S. | At 24 hours following the C/S, the patient will rate her pain, degree of nausea, and itching with verbal numeric rating scales.PCA will also be queried for morphine usage.

SECONDARY OUTCOMES:
A secondary objective is to define the incidence and severity of hydromorphone's side effects. | At 4, 8, 12 and 24 hours following the C/S, the patient will rate her degree of nausea, and itching with verbal numeric rating scales.
A secondary objective is to determine the duration of analgesia | At 24 hours following the C/S, the PCA will be queried for morphine usage.

CONTACTS AND LOCATIONS:
Overall Officials: H.Jane Huffnagle, DO, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] 1. Dixon WJ, Massey FJ. Introduction to statistical analysis. 4th ed. New York: McGraw-Hill, 1983; 377-441. 2. Dixon WJ. Staircase bioassay: the up-and-down method. Neurosci Biobehav Rev 1991;15:47-50. 3. AANA J. 2012 Aug;80(4 Suppl):S25-32. 4. AANA J. 2011 Oct;79(5):427-32. 5. Abram SE, Mampilly GA, Milosavljevic D. Anesthesiology 1997;87:127-134. 6. Drakeford MK, Pettine KA, Brookshire L, Ebert F. J Bone Joint Surg Am. 1991;73:424-428. 7. Rathmell JP, Lair TR, Nauman B. Anesth Analg 2005;101(suppl 5):30-43. 8. Sinatra RS, deLeon-Casasola OA, Ginsberg B, Viscusi ER, editors. Acute Pain Management, chapter 16, pp232. 9. Gautier P, Vandepitte C, Ramquet C., et al. Anesth Analg 2011;113:951-55. 10. O'Donnell DB, Iohom G. Anesthesiology 2009;111:25-9. 11. Vandepitte C, Gautier P, Xu D, et al. Anesthesiology 2013;118:863-7